CLINICAL TRIAL: NCT02740634
Title: Molecular and Structural Imaging in Alzheimer's Disease: A Longitudinal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer Whitwell, Associate Professor of Radiology, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-008682; R01AG050603 (NIH)
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Atypical Alzheimer's Disease; Logopenic Progressive Aphasia (LPA); Posterior Cortical Atrophy (PCA); Alzheimer Disease; Alzheimer Disease, Early Onset; Amnestic Disorder; Amnestic Symptoms; Amnestic Mild Cognitive Disorder
Keywords: PCA; LPA; AD; Amnestic AD
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tau PET Scan, F-18 AV 1451 (Experimental): All subjects will receive two Tau PET scans during this study.
  Interventions: Drug: F-18 AV 1451; Drug: C-11 PiB
- PiB PET Scan, C-11 PiB (Experimental): All subjects will receive two PiB PET scans during this study.
  Interventions: Drug: F-18 AV 1451; Drug: C-11 PiB

INTERVENTIONS:
Drug: F-18 AV 1451 — Tau binding agent
Drug: C-11 PiB — Amyloid binding agent

SUMMARY:
This is a neuroimaging study designed to learn more about amyloid and tau burden in the brain of patients with typical and atypical Alzheimer's Disease and how burden may change over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 21
* Must have an informant who will be able to provide independent evaluation of functioning
* English is primary language
* All subjects must have insidious onset, report progression of their symptoms, and meet current clinical diagnostic criteria for typical amnestic AD or an atypical AD syndrome such as Logopenic Aphasia (LPA) or Posterior Cortical Atrophy (PCA).
* All subjects with Logopenic Aphasia (LPA) must present with early and dominant impairments in language
* All subjects with typical amnestic AD must have relative preservation of episodic memory compared to impairment in the non-episodic memory domain

Exclusion Criteria:

* If you have had a stroke or tumor that could explain your symptoms
* Subjects that present with early episodic memory impairment or meet clinical criteria for mild cognitive impairment will not be recruited into the study
* Subjects that meet specific criteria for another neurodegenerative disorder, including behavioral variant frontotemporal dementia, semantic dementia, primary progressive apraxia of speech, probable corticobasal syndrome, or progressive supranuclear palsy, will be excluded
* Subjects will be excluded if they have poor vision (20/400)
* Women that are pregnant or post-partum and breast-feeding will be excluded
* Subjects will be excluded from the study if they are unable to undergo the tau-PET scan due to a prolonged QT interval on ECG, or if they have any of the following genetic conditions which can increase the chance of cancer: Cowden disease, Lynch syndrome, hypogammaglobulinemia, Wiskott-Aldrich syndrome, and Down's syndrome
* Subjects will also be excluded if MRI is contraindicated (metal in head, cardiac pace maker, e.t.c.), if there is severe claustrophobia, if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma or intracranial neoplasm), or if they are medically unstable or are on medications that might affect brain structure or metabolism,(e.g. chemotherapy)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Amount of Amyloid protein in the brain of patients with Logopenic Aphasia (LPA) or Posterior Cortical Atrophy (PCA). | 5 years
Amount of Tau protein in the brain of patients with Logopenic Aphasia (LPA) or Posterior Cortical Atrophy (PCA). | 5 years

SECONDARY OUTCOMES:
Rates of change in amyloid-PET burden over time. | baseline, 1 year
Rates of change in tau-PET burden over time. | baseline, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Whitwell, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials